CLINICAL TRIAL: NCT05649254
Title: Immediate Effect of Transcutaneous Electrical Nerve Stimulation on Muscle Tone in Children With Spastic Cerebral Palsy
Brief Title: Effect of TENS in Children With Spastic Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amgad Elwy Ali Hussein, Principal Investigator, Cairo University
Other Study IDs: TENS IN CP CHILDREN
Record Dates: First submitted 2022-11-21; First posted 2022-12-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: TENS
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: in which TENS application will be applied
- Control group: placebo treatment

SUMMARY:
TENS is cheap and simple tool for physiotherapist, free of many side effects compared with other tools. so The aim of study was record the effect of TENS on calf muscle tone in spastic cerebral palsy children.

DETAILED DESCRIPTION:
The Significance of this study is to determine whether TENS could have an immediate effect on reduction of spasticity in children diagnosed with spastic cerebral palsy by studying the change of spasticity of ankle plantarflexors immediately after applying TENS to the ankle dorsiflexors.

Muscle tone assessment will be applied before and after the application using objective tool which is electromyography and subjectively by using modified Ashworth scale and goniometer, to be insured is there is an immediate effect of TENS on muscle tone of calf muscle or not.

ELIGIBILITY:
Inclusion Criteria:

* The children will be included in this study is according to the following criteria

  1. Cerebral palsy spastic diaplegia.
  2. Their age ranged from 3-10 years.
  3. Both Sexes were included.
  4. The subjects with mild to moderate muscle tone according to MAS in which mild is 1 and 1+ , and moderate is 2.

Exclusion Criteria:

* The subject will be excluded if he/she has one or more of the following criteria:

  1. Children with a history of seizures.
  2. Children who could not lie prone for any cause.
  3. Children who could not react to pain.
  4. Children who had applied any surgical procedure which affect muscle tone or any inhibitory injections like BOTOX.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children diagnosed with spastic cerebral palsy diplgeia of both sexes will be selected from El-Menshawy public governmental hospital in Tanta City following the official rules and after gaining the agreements of the parents and explaining the aim and procedures of the study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
MUSCLE TONE that will be measured subjectively by modified ashwoth scale | Baseline
  the study will assess if TENS have effect on muscle tone or not the tone will be measured subjectivly by using modified ashworth scale . The Modified Ashworth scale evaluation involves the rater manually moving a limb through the range of motion to passively stretch specific muscle groups and a six-point ordinal scale for grading the resistance encountered during such passive muscle stretching. MAS grades of spasticity are as follows: 0 = normal muscle tone; 1=slight increase in muscle tone, manifested by catch and release or by minimal resistance at the end; 1+=slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout; 2=more marked increase in muscle tone, but limb easily flexed; 3=considerable increase in muscle tone, passive movement difficult; and 4 = limb rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Osama Sayed, Phd, Study Director — Assistant Professor at Cairo university
Locations (1):
- Faculty of physical therapy Cairo university, Giza, Dokki, Egypt

REFERENCES:
- [Background] Mills PB, Dossa F. Transcutaneous Electrical Nerve Stimulation for Management of Limb Spasticity: A Systematic Review. Am J Phys Med Rehabil. 2016 Apr;95(4):309-18. doi: 10.1097/PHM.0000000000000437. PMID 26829077
- [Result] Aydin G, Tomruk S, Keles I, Demir SO, Orkun S. Transcutaneous electrical nerve stimulation versus baclofen in spasticity: clinical and electrophysiologic comparison. Am J Phys Med Rehabil. 2005 Aug;84(8):584-92. doi: 10.1097/01.phm.0000171173.86312.69. PMID 16034227